CLINICAL TRIAL: NCT05954637
Title: Correlation of Structure and Function in Glaucoma
Status: Completed | Type: Observational
Sponsor: Vienna Hospital Association (Other Government)
Responsible Party: Principal Investigator, Prim. Univ.-Prof. Dr. Pia Veronika Vécsei-Marlovits, MSc, MB, Head of Department of Ophthalmology, Vienna Hospital Association
Other Study IDs: struct_funct_glaucoma
Record Dates: First submitted 2023-07-10; First posted 2023-07-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Optical coherence tomography — Heidelberg Engineering Spectralis

SUMMARY:
The aim of the study is to correlate structure and function in patients with glaucoma. To this end, a cross-sectional study unsing perimetry and optical coherence tomography is performed.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of glaucomatous optic neuropathy

Exclusion Criteria:

* Age < 18 years
* Diabetes
* Pregnancy
* Hypertensive retinopathy
* Smoking
* Intraocular surgery 1 month prior to study entry
* Systemic or ocular disease, excluding glaucoma, which the investigator believes could affect the test results
* Insufficient quality of the optical coherence tomography imaging
* Insufficient cooperation during examinations or measurements

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Department of Ophthalmology, Clinic Hietzing, Vienna Healthcare Group, who have been diagnosed with "glaucomatous optic neuropathy" are eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Association of retinal sensitivity with peripapillary retinal nerve fiber layer thickness | 1 day
Association of retinal sensitivity with peripapillary vessel density | 1 day

SECONDARY OUTCOMES:
Glaucoma Activity Limitation score | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pia V Vécsei-Marlovits, MD, MSc, MBA, Principal Investigator — Department of Ophthalmology, Clinic Hietzing, Vienna Healthcare Group
Locations (1):
- Department of Ophthalmology, Clinic Hietzing, Vienna Healthcare Group, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided